CLINICAL TRIAL: NCT01289704
Title: A Multicenter Study to Evaluate the Effects on Charcot-Marie-Tooth Neuropathy Type 1A of a Composite Treadmill, Stretching and Proprioceptive Exercise (TreSPE) Rehabilitation Program.
Brief Title: Treadmill, Stretching and Proprioceptive Exercise (TreSPE) Rehabilitation Program for Charcot-Marie-Tooth Neuropathy Type 1A (CMT1A)
Acronym: TreSPE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Responsible Party: Gianluigi Mancardi, Neuroscience, Ophtalmology and Genetic Departement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GUP09013
Record Dates: First submitted 2011-01-24; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2010-10

CONDITIONS: Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth Disease Type 1A
Keywords: Charcot-Marie-Tooth disease,; CMT1A,; rehabilitation,; treadmill,; stretching,; proprioception,; Randomised Controlled Trial.
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TreSPE (Experimental): Treatment with treadmill, proprioceptive and stretching exercises
  Interventions: Other: TreSPE
- SPE (Active Comparator): Proprioceptive and stretching exercises
  Interventions: Other: TreSPE; Other: SPE

INTERVENTIONS:
Other: TreSPE — 1. treadmill: 5'warm up, 20'aerobic exercise (gradually incremented to 30', from session to session, if possible), 5'warm down, controlling hearth rate, blood pressure and SaO2.
  2. Respiratory Physiotherapy: positive Expiratory Pressure (PEP) bottle for 10' (in various postures), and postural training, for the other 10'.
  3. Stretching for 20', of the triceps surae, tibialis posterior, extensor and flexors digitorum longus and brevis, both at the bed and in a static position.
  4. Proprioceptive and postural kinesitherapy according to the Perfetti method.
  5. Balance Exercising consists of exercises carried on by basculating bars with improving difficulties in the instruments utilized and in the tasks with therapist supervision and near a handbar preventing falls.
  Other Names: SPE
Other: SPE — 1. Respiratory Physiotherapy for 20', consisting of Positive Expiratory Pressure (PEP) bottle for 10' (in various postures), and postural training according to the Mèzières technique, for the other 10'.
  2. Stretching for 20', of the triceps surae, tibialis posterior, extensor and flexors longus and brevis, both at the bed and in a static position.
  3. Proprioceptive and postural kinesitherapy according to the neurocognitive method.
  4. Balance Exercising consists of exercises carried on by moving bars with improving difficulties in the instruments utilized and in the tasks with therapist supervision and near a handlebar preventing falls.
  Arms: SPE

SUMMARY:
Charcot-Marie-Tooth neuropathy type 1A (CMT1A) is one of the most common inherited neurological disorders. The study will evaluate the efficacy and safety of an innovative rehabilitation protocol constituted by exercises at the treadmill and by a stretching and proprioceptive approach. A total of 92 patients will be enrolled in the study and treated in a controlled, randomized, single blind, way. To recruit a high number of patients with CMT1A the study will be multicentric and will comprehend four of the most active clinical centers in the field of CMT, in Italy. People with CMT1A are very motivated in entering rehabilitation protocols because to date there is no effective therapy for this disease. Therefore, the investigators expect a high compliance by the patients. With the present project the investigators plan to clarify several unanswered questions: 1) the efficacy and safety of treadmill over a more conventional protocol; 2) the duration and frequency of any rehabilitation treatment; 3) the most sensitive outcome measures to evaluate the efficacy of rehabilitation approach in patients with CMT.

DETAILED DESCRIPTION:
A multicentre, prospective, randomised, controlled, single blind study to evaluate the impact of aerobic exercise, based on a tightly controlled program at the treadmill, on the rehabilitation therapy of CMT 1A neuropathy.

Comparing aerobic training at the treadmill combined with respiratory physiotherapy, stretching and proprioceptive exercises (TreSPE- treated group) with a more conventional treatment only composed by respiratory physiotherapy, stretching and proprioceptive exercises (SPE- control group) will provide information on the impact of Treadmill in CMT1A.

92 patients (23 per centre) will be enrolled and randomly assigned to TreSPE (n = 46) or to SPE (n = 46). Both groups will be treated for three months and followed up for six months.

No serious side effects are expected with TreSPE, as also suggested by our preliminary results. For safety reasons blood pressure (BP), heart rate (HR) and an electrocardiogram will be recorded during the rehabilitation treatment when the treating physician considers it necessary. The patients will be allowed, if needed, to hold at the parallel bars of the treadmill during exercise. According to the American Thoracic Society (ATS) guidelines the cardiopulmonary exercise test will be interrupted if BP raises at 240/120 and/or HR to 220-patients age.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CMT1A
* Genetic confirmation (17p112 chromosome duplication)
* Age 18 - 70 years old
* Ability to accomplish the primary outcome measure (10 meter walking test) without support, with or without ankle foot orthoses (AFO)
* Ability to walk on a treadmill on a horizontal plane for 20 minutes at a speed of 1.5 km/h with or without support at the bars
* Score at the Mobility Scale between 2 and 11
* Signed written informed consent to participate

Exclusion Criteria:

* Diagnosis of Hereditary Neuropathy with Liability to Pressure Palsies (HNPP) or any other type of CMT
* Other associated causes of neuropathy
* Vestibular affections, psychiatric, cardiovascular and lung disorders or severe arthropathic changes in the lower limbs
* Non ambulating patients or patients always requiring even monolateral support to walk
* Other neurological disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Walking ability of patients will be evaluated as the time needed to walk for 10 meters at normal speed for the patients | Baseline: 1 day before the rehabilitative protocol starts (T1)
  The walking ability of patients will be evaluated through the "10 meters timed walk test" which will be performed at baseline (T1 or day-1), at the end of the three months of treatment (T2 or day90) and at the end of the three months of follow up (T3 or day180).
Walking ability of patients will be evaluated after finishing the treatment as the time needed to walk for 10 meters at normal speed for the patients | at the end of treatment: day 90 (T2)
  The walking ability of patients will be evaluated through the "10 meters timed walk test" which will be performed at baseline (T1 or day-1), at the end of the three months of treatment (T2 or day90) and at the end of the three months of follow up (T3 or day180).
Walking ability of patients will be evaluated after finishing the treatment as the time needed to walk for 10 meters at normal speed for the patients | at the end of follow up: day 180 (T3)
  The walking ability of patients will be evaluated through the "10 meters timed walk test" which will be performed at baseline (T1 or day-1), at the end of the three months of treatment (T2 or day90) and at the end of the three months of follow up (T3 or day180).

SECONDARY OUTCOMES:
Balance will be evaluated through the Berg Scale | Baseline: 1 day before the rehabilitative protocol starts
  The Berg scale is a tool to evaluate balance and ranges from 0 to 36 points being 36 normal
Balance will be evaluated through the Berg Scale | at the end of treatment: day 90 (T2)
  The Berg scale is a tool to evaluate balance and ranges from 0 to 36 points being 36 normal
balance will be evaluted through the Berg scale | at the end of follow up: day 180 (T3)
  The Berg scale is a tool to evaluate balance and ranges from 0 to 36 points being 36 normal
Quality of life will be evaluated through the SF - 36 questionnaire | Baseline: 1 day before the rehabilitative protocol starts (T1)
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Quality of life will be evaluated through the SF - 36 questionnaire | at the end of treatment: day 90 (T2)
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Quality of life will be evaluated through the SF - 36 questionnaire | at the end of follow up: day 180 (T3)
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo E Schenone, MD, Principal Investigator — University of Genova
Locations (4):
- Italy (4):
  - University of Genoa, Genoa
  - I.R.C.C.S. Foundation, Besta Institute, Milan
  - Don Carlo Gnocchi Foundation, Rome
  - Departement of Neurological and Visual Sciences, University of Verona, Verona

REFERENCES:
- [Background] Grandis M, Shy ME. Current Therapy for Charcot-Marie-Tooth Disease. Curr Treat Options Neurol. 2005 Jan;7(1):23-31. doi: 10.1007/s11940-005-0003-5. PMID 15610704
- [Background] Young P, De Jonghe P, Stogbauer F, Butterfass-Bahloul T. Treatment for Charcot-Marie-Tooth disease. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD006052. doi: 10.1002/14651858.CD006052.pub2. PMID 18254090
- [Background] Passage E, Norreel JC, Noack-Fraissignes P, Sanguedolce V, Pizant J, Thirion X, Robaglia-Schlupp A, Pellissier JF, Fontes M. Ascorbic acid treatment corrects the phenotype of a mouse model of Charcot-Marie-Tooth disease. Nat Med. 2004 Apr;10(4):396-401. doi: 10.1038/nm1023. Epub 2004 Mar 21. PMID 15034573
- [Background] Pareyson D, Schenone A, Fabrizi GM, Santoro L, Padua L, Quattrone A, Vita G, Gemignani F, Visioli F, Solari A; CMT-TRIAAL Group. A multicenter, randomized, double-blind, placebo-controlled trial of long-term ascorbic acid treatment in Charcot-Marie-Tooth disease type 1A (CMT-TRIAAL): the study protocol [EudraCT no.: 2006-000032-27]. Pharmacol Res. 2006 Dec;54(6):436-41. doi: 10.1016/j.phrs.2006.09.001. Epub 2006 Sep 9. PMID 17029975
- [Background] Carter GT, Han JJ, Mayadev A, Weiss MD. Modafinil reduces fatigue in Charcot-Marie-Tooth disease type 1A: a case series. Am J Hosp Palliat Care. 2006 Oct-Nov;23(5):412-6. doi: 10.1177/1049909106292169. PMID 17060310
- [Background] Aitkens SG, McCrory MA, Kilmer DD, Bernauer EM. Moderate resistance exercise program: its effect in slowly progressive neuromuscular disease. Arch Phys Med Rehabil. 1993 Jul;74(7):711-5. doi: 10.1016/0003-9993(93)90031-5. PMID 8328892
- [Background] Kilmer DD, McCrory MA, Wright NC, Aitkens SG, Bernauer EM. The effect of a high resistance exercise program in slowly progressive neuromuscular disease. Arch Phys Med Rehabil. 1994 May;75(5):560-3. PMID 8185450
- [Background] van Pomeren M, Selles RW, van Ginneken BT, Schreuders TA, Janssen WG, Stam HJ. The hypothesis of overwork weakness in Charcot-Marie-Tooth: a critical evaluation. J Rehabil Med. 2009 Jan;41(1):32-4. doi: 10.2340/16501977-0274. PMID 19197566
- [Background] Carter GT, Abresch RT, Fowler WM Jr, Johnson ER, Kilmer DD, McDonald CM. Profiles of neuromuscular diseases. Hereditary motor and sensory neuropathy, types I and II. Am J Phys Med Rehabil. 1995 Sep-Oct;74(5 Suppl):S140-9. doi: 10.1097/00002060-199509001-00008. PMID 7576421
- [Background] Carter GT, Kilmer DD, Bonekat HW, Lieberman JS, Fowler WM Jr. Evaluation of phrenic nerve and pulmonary function in hereditary motor and sensory neuropathy, type I. Muscle Nerve. 1992 Apr;15(4):459-62. doi: 10.1002/mus.880150407. PMID 1565114
- [Background] Sackley C, Disler PB, Turner-Stokes L, Wade DT. Rehabilitation interventions for foot drop in neuromuscular disease. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD003908. doi: 10.1002/14651858.CD003908.pub2. PMID 17443532
- [Background] Solari A, Laura M, Salsano E, Radice D, Pareyson D; CMT-TRIAAL Study Group. Reliability of clinical outcome measures in Charcot-Marie-Tooth disease. Neuromuscul Disord. 2008 Jan;18(1):19-26. doi: 10.1016/j.nmd.2007.09.006. Epub 2007 Oct 26. PMID 17964785
- [Background] Florence JM, Hagberg JM. Effect of training on the exercise responses of neuromuscular disease patients. Med Sci Sports Exerc. 1984 Oct;16(5):460-5. doi: 10.1249/00005768-198410000-00007. PMID 6513764
- [Background] Jones DR, Speier J, Canine K, Owen R, Stull GA. Cardiorespiratory responses to aerobic training by patients with postpoliomyelitis sequelae. JAMA. 1989 Jun 9;261(22):3255-8. PMID 2654435
- [Background] Aitkens S, Kilmer DD, Wright NC, McCrory MA. Metabolic syndrome in neuromuscular disease. Arch Phys Med Rehabil. 2005 May;86(5):1030-6. doi: 10.1016/j.apmr.2004.09.012. PMID 15895353
- [Background] Pfeiffer G, Wicklein EM, Ratusinski T, Schmitt L, Kunze K. Disability and quality of life in Charcot-Marie-Tooth disease type 1. J Neurol Neurosurg Psychiatry. 2001 Apr;70(4):548-50. doi: 10.1136/jnnp.70.4.548. PMID 11254787
- [Background] Vinci P, Serrao M, Millul A, Deidda A, De Santis F, Capici S, Martini D, Pierelli F, Santilli V. Quality of life in patients with Charcot-Marie-Tooth disease. Neurology. 2005 Sep 27;65(6):922-4. doi: 10.1212/01.wnl.0000176062.44360.49. PMID 16186535
- [Background] Shy ME, Blake J, Krajewski K, Fuerst DR, Laura M, Hahn AF, Li J, Lewis RA, Reilly M. Reliability and validity of the CMT neuropathy score as a measure of disability. Neurology. 2005 Apr 12;64(7):1209-14. doi: 10.1212/01.WNL.0000156517.00615.A3. PMID 15824348
- [Background] Graham RC, Hughes RA. Clinimetric properties of a walking scale in peripheral neuropathy. J Neurol Neurosurg Psychiatry. 2006 Aug;77(8):977-9. doi: 10.1136/jnnp.2005.081497. Epub 2006 Mar 30. PMID 16574732
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547
- See also: Acmt-Rete is a non-profit organization made by a group of patients to help the CMT community and to promote research in the field of hereditary neuropathies — http://www.acmt-rete.it